CLINICAL TRIAL: NCT01127516
Title: The Causes and Interpretation of Low-level Resistance in Staphylococcus Aureus to Vancomycin Among a Network of Academic Medical Center Hospitals
Brief Title: The Causes and Interpretation of Low-level Resistance in Staphylococcus Aureus
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: PT105051
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Staphylococcus Aureus
Keywords: Susceptibility testing; Antimicrobial stewardship
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The hypothesis of this investigation is that rate of isolation of resistant nosocomial pathogens can be explained by a combination of measures that include, among other things, antimicrobial drug use, infection control efforts, patient mix and antimicrobial stewardship efforts. The short term goal of this investigation is to improve our understanding of the relationships between antimicrobial stewardship program efforts (and actual antimicrobial drug use), and infection control efforts to the incidence rates of MSSA, MRSA, h-VISA and SA-MICcreep. The long term goal of this investigation is to design interventions that will improve antimicrobial drug use and decrease cross-transmission of resistant bacteria, resulting in a decrease in the rates of infection caused resistant hospital organisms.

DETAILED DESCRIPTION:
Study Design

We propose to survey clinical pharmacists, infectious diseases practitioners and clinical microbiologists at these 53 hospitals during the summer of 2009 to characterize the hospital policy toward isolation of SA-MICcreep and to investigate the relationship of SA-MICcreep to vancomycin use. Specifically, we will determine (1) if the hospital attempts to isolate SA-MICcreep (2) the method(s) of testing SA susceptibility to vancomycin, (3) interpretative criteria for MICs to vancomycin and whether there is a policy toward differential treatment of isolated with SA-MICcreep. In addition we will determine (1) the relationship of SA-MICcreep to vancomycin use and (2) the relationship to other hospital and patient demographics to SA-MICcreep. A pilot study (Dec. 2008) found that 7 of 8 hospitals surveyed do determine the vancomycin MIC for Staphylococcus aureus. However the interpretation of these findings, and the action taken, differ between hospitals. This may be because this is a newly described phenomenon, and professional organizations have not yet issued guidelines regarding the interpretation of these isolates (6).

We have measured vancomycin use by the following methods at each hospital:

* Days of therapy/1000 patient days.
* Mean duration of vancomycin therapy (days).
* Proportion of adult patients who receive vancomycin (%).
* Vancomycin "Intensity Index": The product of #2 and #3.

We will also measure the use of other antibacterial drugs that are used to treat infections caused by Staphylococcus aureus including linezolid and daptomycin as these drugs may reduce the isolation of SA-MICcreep.

The survey instrument will include requests for the following information:

1. Does the clinical microbiology laboratory make an attempt to identify MIC creep for clinical isolates of Staphylococcus aureus?

1. If yes, when did this policy begin?
2. Are all Staphylococcus aureus isolates tested (i.e., MSSA and MRSA) or only MRSA?
3. Are all clinical isolated routinely tested, or only selected isolates (e.g., only by request from ID, or only blood isolates, or only isolates from ICU patients, etc.)
4. What method(s) is used to determine the MIC to vancomycin?
5. What MIC is thought to warrant concern? (e.g., 1.0, 1.5, 2.0 mcg/ml) ?
6. What action, if any, is taken as a function of the MIC to vancomycin?
7. Is "more aggressive" therapy with vancomycin attempted if an isolate of concern is identified, or is alternative therapy recommended or routinely implemented?
8. If alternative therapy is routinely administered, what is that therapy?

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients

Exclusion Criteria:

* Pediatric inpatients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult inpatients
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Proportion of hospitals that test for MIC creep to vancomycin | 2009
  Survey of hospitals participating in the UHC consortium

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Commonwealth University School ofPharamcy, Richmond, Virginia, United States